CLINICAL TRIAL: NCT06581380
Title: A Multicenter, Randomized, Positive-Controlled, Open-label, Phase 3 Study of JK-1201I Compared with Topotecan in Patients with Relapsed Extensive Stage Small Cell Lung Cancer After Platinum-based First-line Chemotherapy
Brief Title: JK-1201I Compared with Topotecan in Patients with Relapsed Extensive Stage Small Cell Lung Cancer
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: JenKem Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JK-1201I-301
Record Dates: First submitted 2024-08-29; First posted 2024-09-03 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- JK-1201I (Experimental): Participants will receive JK-1201I as an intravenous (IV) infusion at dose of 180mg/m2 on Day 1 of each 21-day cycle until a treatment discontinuation criterion is met as specified in the protocol.
  Interventions: Drug: JK-1201I
- Topotecan (Active Comparator): Participants will receive topotecan until a treatment discontinuation criterion is met as specified in the protocol.
  Interventions: Drug: Topotecan

INTERVENTIONS:
Drug: JK-1201I — JK-1201I will be administered as an IV infusion at dose of 180mg/m2 on Day 1 of each 21-day cycle.
  Arms: JK-1201I
Drug: Topotecan — Topotecan will be administered per drug label.
  Arms: Topotecan

SUMMARY:
This study was designed to compare the efficacy and safety of JK-1201I with Topotecan in patients with relapsed extensive stage small cell lung cancer (ES SCLC).

DETAILED DESCRIPTION:
This is a multicenter, randomized, positive-controlled, open-label, phase 3 study comparing JK-1201I with topotecan in patients with Relapsed Extensive Stage Small Cell Lung Cancer that had relapsed or disease progression on or after platinum-based first-line chemotherapy.

Patients will be randomized by a ratio of 1:1 to receive JK-1201I or topotecan until disease progression.

of JK-1201I Compared with Topotecan in Patients With Relapsed Extensive Stage Small Cell Lung Cancer After Platinum-based First-line Chemotherapy The primary objective of this study is to assess whether treatment with JK-1201I prolongs overall survival (OS) compared with treatment of topotecan among patients with relapsed ES SCLC.

The secondary objectives of the study are to further evaluate the efficacy, safety and population pharmacokinetics of JK-1201I.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all the following criteria to be eligible for randomization into the study:

1. Sign and date the informed consent form prior to the start of any study-specific qualification procedures.
2. Male or female aged ≥18 years and ≤70 years.
3. Histologically or cytologically documented SCLC.
4. Has received prior therapy with only one prior platinum-based line as systemic therapy for ES SCLC and Disease progression on or after first-line platinum-based regimens (≤ 6 months).
5. Has at least 1 measurable lesion according to RECIST v1.1.
6. Has ECOG PS of ≤1.

Exclusion Criteria:

Participants who meet any of the following criteria will be disqualified from entering the study:

1. Hypersensitivity to any ingredient of JK-1201I and Topotecan.
2. Has received prior treatment with DNA topoisomerase I inhibitor agents.
3. Has received prior therapy with ≥2 line as systemic therapy for extensive-stage SCLC.
4. Chemotherapy-free interval within 4 weeks before the first use of the study drug. Radiotherapy with a limited field of radiation for palliation within 2 weeks before the first use of the study drug. Used biotherapy drugs within 2 weeks before the first use of the study drug.
5. Severe gastrointestinal illnesses as defined in the protocol within 6 months before the first use of the study drug.
6. Local symptoms of tumors requiring radiotherapy or surgical treatment as defined in the protocol.
7. Untreated or symptomatic brain metastases with exceptions defined in the protocol.
8. Severe pulmonary illnesses within 6 months before the first use of the study drug.
9. Uncontrolled hydrothorax and ascites.
10. Unresolved toxicity from prior anti-tumor therapy, defined as not having resolved to Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 grade 1 with exceptions defined in the protocol.
11. Severe infections within 4 weeks before the first use of the study drug.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 394 (Estimated)
Dates: Start 2024-09-16 (Estimated); Primary Completion 2027-11-16 (Estimated); Study Completion 2028-04-16 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | From the date of randomization to the date of death due to any cause; Up to approximately 3.5 years.
  Overall survival is defined as the time interval from randomization to death due to any cause.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) Assessed by Independent Response Evaluation Committee (IREC) and Investigators | From the date of randomization to documented progressive disease, death, lost to follow-up, or withdrawal by the participant; Up to approximately 3.5 years.
  Confirmed ORR is defined as the proportion of participants who have achieved a best overall response of confirmed complete response (CR), confirmed partial response (PR) per IREC and investigator per Response Evaluation Criteria In Solid Tumors (RECIST) v1.1.
Disease Control Rate (DCR) Assessed by Independent Response Evaluation Committee (IREC) and Investigators | From the date of randomization to documented progressive disease, death, lost to follow-up, or withdrawal by the participant; Up to approximately 3.5 years.
  Disease control rate is defined as the proportion of participants who have achieved a best overall response of confirmed CR, confirmed PR, or SD (or non-CR/non-PD) per IREC and investigator per Response Evaluation Criteria In Solid Tumors (RECIST) v1.1.
Duration of Response (DoR) Assessed by Independent Response Evaluation Committee (IREC) and Investigators | From the date of first documentation of confirmed response (CR or PR) to the first documentation of progressive disease or death due to any cause, whichever occurs first; Up to approximately 3.5 years.
  Duration of response (DoR) is defined as the time from the date of the first documentation of objective response (complete response [CR] or partial response [PR]) to the date of the first documentation of progressive disease (PD) or death.
Progression-free Survival (PFS) Assessed by Independent Response Evaluation Committee (IREC) and Investigators | From the date of randomization to documented progressive disease, death, lost to follow-up, or withdrawal by the participant; Up to approximately 3.5 years.
  Progression-free Survival (PFS) is defined as the time interval from the randomization to disease progression as per Independent Response Evaluation Committee (IREC) and Investigators assessment or death due to any cause.
Incidence and Grade of Participants with Adverse Events (AE) | From the date of first dose to the end of safety follow-up; Up to approximately 3.5 years
  Adverse Events (AEs) are assessed based on NCI CTCAE v5.0.
Pharmacokinetic Parameter Area Under the Plasma Concentration-Time Curve for JK-1201I, Irinotecan, SN38 and SN38G | Cycle 1 before infusion, and 12, 168, and 240 hours (hrs) post dose; every 2 cycles before infusion, and 12 hrs post dose thereafter up to 3.5 years (each cycle is 21 days)
  Area under the plasma concentration-time curve up to the last quantifiable time point (AUClast) and area under the plasma concentration-time curve dosing interval (AUCtau) will be assessed using Non-linear mixed effect modeling in 80 participants randomized to JK-1201 group.
Pharmacokinetic Parameter Maximum Concentration for JK-1201I, Irinotecan, SN38 and SN38G | Cycle 1 before infusion, and 12, 168, and 240 hours (hrs) post dose; every 2 cycles before infusion, and 12 hrs post dose thereafter up to 3.5 years (each cycle is 21 days)
  Maximum concentration (Cmax) will be assessed using Non-linear mixed effect modeling in 80 participants randomized to JK-1201 group.

IPD SHARING:
Plan to Share IPD: Undecided